CLINICAL TRIAL: NCT00748007
Title: Efficacy of Rivastigmine in Patients With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Wuh-Liang Hwu, National Taiwan University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200709028M
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Down Syndrome
Keywords: Down syndrome, cholinesterase inhibitor, Rivastigmine
MeSH Terms: conditions — Down Syndrome | interventions — Rivastigmine; Cholinesterase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Rivastigmine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine — Exelon (1.5mg/cap) 1.5 mg bid
  Other Names: Exelon and placebo; Cholinesterase inhibitor

SUMMARY:
This study is to understand the efficacy on language and cognitive function in Down syndrome patients who take Rivastigmine.

DETAILED DESCRIPTION:
Down syndrome (DS) is the most common cause of mental retardation due to chromosome anomaly. Besides defects in cognition, DS patients after 30 yeas old will have early dementia. Etiology of early dementia is known to be related with APP gene dosage triplication that is similar to the neuropathological change in Alzheimer disease (AD). It has been known that the cognitive degeneration in AD is related with decrement of cholinergic neurons in the brain. And the clinical improvement or delay in degeneration of cognitive function after utilization of cholinesterase inhibitor had been observed in mild to moderate AD patients. In DS brain, it has been also noted to be lower acetylcholine, supporting the relationship of pathology between DS and AD. Since 1999, Kishnani et al started to treat adult DS patients with cholinesterase inhibitor (Donepezil). Data showed the improvement of cognition and life quality in DS patients with dementia. Recently, data showed the low cholinergic neuron in DS brain might be a cause of cognitive dysfunction in DS. Therefore, early treatment of cholinesterase inhibitor in DS patients had been proposed to alleviate cognitive dysfunction. Since 2004, Kishnani et al started to treat DS children with Donepezil and Rivastigmine. Some patients showed improvement of language ability, memory, and attention. We are going to conduct a randomized, double-blind, placebo-controlled, crossover design, 12-month trial. Subjects who are enrolled in this study will be randomized into two groups. Each group will receive Rivastigmine and placebo in different order for 6 months. Neuropsychological assessment including Vineland Adaptive Behavior Scales and NEPSY will be evaluated before and after medication. Through this, we wish to understand the efficacy of this drug in the role of improving cognitive functioning in our patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 8 years old
2. Diagnosed to have Down syndrome.
3. Full IQ > 40
4. Patients and caregiver agreed and could participated in this trial
5. Have to sign permit. If patient is less than 18 years old, inform consent should be singed by parents

Exclusion Criteria:

1. Known to be allergy to Rivastigmine
2. Currently uncontrolled heart, gastrointestinal, renal or central nervous system problems that could effect evaluation or compliance A. Heart rate less than 50/min B. Patients has uncontrolled severe disease such as gastric ulcer, uncontrolled hypothyroidism, vit B12 deficiency, severe renal or liver disease, diabetes, or asthma C. Uncontrolled psychiatric disease D. Diagnosed to have primary neurodegenerative disease such as Huntington's disease, uncontrolled seizure, delirium E. Hearing defects or vision effect that will affect neuropsychiatric evaluations F. Pregnancy
3. Currently usage of special medications A. Toxic agents to major organs 4 weeks before using Rivastigmine B. Taking drugs for psychiatric problems 4 weeks before using Rivastigmine C. Taking Rivastigmine 6 weeks before entering the trial D. Taking other acetylcholinesterase inhibitors such as Donepezil (Aricept)、Galantamine (Razadyne, Razadyne ER)、Anticholinergic agents, such as diphenhydramine (Benadryl), oxybutynin (Ditropan), or N-Methyl-D-Aspartate (NMDA) receptor antagonist such as Memantine (Namenda)
4. Not willing to cooperate with follow up programs
5. Other conditions that doctors or investigators consider not suitable to enter this trial

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Scores of Vineland Adaptive Behavior Scales (VABS), Scores of WISC digit span, Scores of Leiter-R Forward memory , Scores of PPVT, | at 24, and 54 weeks

SECONDARY OUTCOMES:
Scores of NEPSY test for Visuospatial and Design Coping, Scores of Visuomotor Precision, Scores of WPPSI Sentences, Scores of Score for Character Recognitions by School Grade, and Scores of Test for Mathematic Ability for Children | 24 and 54 wks

CONTACTS AND LOCATIONS:
Overall Officials: Wuh-Liang Hwu, MD. PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Medical Genetics, National Taiwan University Hospital, Taipei, Taiwan